CLINICAL TRIAL: NCT02391402
Title: Cognitively Augmented Behavioral Activation for Veterans With Comorbid TBI/PTSD
Acronym: CABA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1189-I
Record Dates: First submitted 2015-02-17; First posted 2015-03-18 (Estimated); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-04

CONDITIONS: Traumatic Brain Injury; Posttraumatic Stress Disorder
Keywords: Brain injury; TBI; PTSD; Polytrauma
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic; Brain Injuries; Multiple Trauma | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CABA (Experimental): CABA uses Behavioral Activation (BA) to identify meaningful goals and activities while learning cognitive skills to aid in working toward those goals. Early sessions of CABA focus on learning about mTBI, PTSD, and lifestyle skills that can improve thinking abilities and mood. Cognitive skills taught each week include internal and external skills to help manage problems with memory, attention, and regulation of thinking processes. Investigators and patients will spend a part of each session applying the cognitive skills to managing real life situations and getting patients active in the service of personal goals.
  Interventions: Behavioral: Cognitively Augmented Behavioral Activation
- TAU (Placebo Comparator): Treatment as Usual (TAU) is the usual care that patients would normally receive at the VA. TAU care involves psychotherapy (counseling) provided by a specialist in the treatment of PTSD. Patients will be offered individual appointments with an experienced provider on the PTSD Clinical Team (PCT). Beyond this, the specific approach will be determined by the patient and his/her provider and may include skills for managing PTSD and/or a chance for the patient to "process" his/her traumatic experiences. Additional treatments may be offered to patients, such as group classes and medications. TAU care may also include additional evaluation and/or treatment of mTBI, provided by the usual care offered in Portland or Seattle's respective neuropsychology clinics. Treatment for mTBI includes individual or group sessions, and is based on clinical need.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Cognitively Augmented Behavioral Activation — CABA uses Behavioral Activation (BA) to identify meaningful goals and activities while learning cognitive skills to aid in working toward those goals. Early sessions of CABA focus on learning about mTBI, PTSD, and lifestyle skills that can improve thinking abilities and mood. Cognitive skills taught each week include internal and external skills to help manage problems with memory, attention, and regulation of thinking processes. Investigators and patients will spend a part of each session applying the cognitive skills to managing real life situations and getting patients active in the service of personal goals.
  Other Names: CABA
  Arms: CABA
Behavioral: Treatment as Usual — TAU care involves psychotherapy (counseling) provided by a specialist in the treatment of PTSD. Patients will be offered individual appointments with an experienced provider on the PTSD Clinical Team (PCT). Beyond this, the specific approach will be determined by the patient and his/her provider and may include skills for managing PTSD and/or a chance for the patient to "process" his/her traumatic experiences. Additional treatments may be offered to patients, such as group classes and medications. TAU care may also include additional evaluation and/or treatment of mTBI, provided by the usual care offered in Portland or Seattle's respective neuropsychology clinics. Treatment for mTBI includes individual or group sessions, and is based on clinical need.
  Other Names: TAU
  Arms: TAU

SUMMARY:
The primary objective of this study is to evaluate the efficacy of Cognitively Augmented Behavioral Activation (CABA), a new hybrid treatment for Veterans diagnosed with comorbid mild Traumatic Brain Injury (mTBI) and posttraumatic stress disorder (PTSD). The study's specific goals are to determine whether: 1) CABA reduces PTSD symptoms in Veterans with mTBI/PTSD, 2) CABA reduces cognitive-related functional impairment in Veterans with mTBI/PTSD, 3) CABA results in improvements in depression symptoms, cognitive functioning, and quality of life in Veterans with mTBI/PTSD; and 4) CABA is an acceptable treatment for Veterans with mTBI/PTSD. The overall goal is to develop an evidence-based manualized treatment for comorbid mTBI/PTSD that can be readily implemented in Veterans Health Administration (VHA) treatment settings.

DETAILED DESCRIPTION:
Veterans historically exhibit high rates of comorbid mTBI/PTSD. Given the comorbidity and neuropsychiatric symptom overlap of these disorders, it can be difficult to determine whether problems and disruptions in functioning are due to mTBI, PTSD, or both. Hence, it is challenging for providers to know how to prioritize these patients' clinical issues and how to effectively treat them. Currently, there are no evidence-based treatments for comorbid mTBI/PTSD. Further, it is unclear to what extent existing treatments for each disorder can be adherently and effectively implemented for the other. As such, most current treatment recommendations suggest a holistic or integrated approach to treatment for comorbid mTBI/PTSD targeting symptoms and functionality rather than underlying etiology. Investigators are proposing a treatment for comorbid mTBI and PTSD that directly targets daily functioning and quality of life.

The study design makes use of the convergent availability of resources at the two participating Veterans Administration Health Care Systems in Portland, Oregon, and Seattle, Washington to conduct a Randomized Controlled Trial (RCT) of CABA. The study will recruit a total of 192 Veterans less than or equal to 55 years of age, 96 participants at each site, enrolled at participating VA Medical Centers (VAMCs) who are diagnosed with both mTBI and PTSD. Eligible participants will be randomly assigned to either the CABA or Treatment as Usual (TAU) group. Participants in the CABA group will receive the CABA intervention during the first 14 weeks of their participation in the study, whereas TAU participants will continue to receive TAU (usual care in a PTSD specialty treatment clinic, but no CABA) during their participation in the study. Both groups will undergo evaluations at baseline, 7 weeks (mid-treatment), 14 weeks (post-treatment), and 39 weeks (6 month follow-up). During their study participation, all participants will continue to receive their usual medical care.

ELIGIBILITY:
Inclusion Criteria:

* Veterans 55 years of age enrolled at participating VA sites able to provide informed consent.
* Diagnosis of PTSD based on the Clinician Administered PTSD Scale.
* Positive screen on the Structured Interview for Collecting Head Trauma Event Characteristics as per the VA/Department of Defense (DoD) Clinical Practice Guideline for Management of Concussion/mTBI; AND endorsed any of the Neurobehavioral Symptom Inventory (NSI) cognitive symptoms items (items 13-17).
* English speaking, able to travel to the primary care clinics weekly for 10 sessions and for the follow-up assessments, and willing to refrain from the initiation of additional mental health treatment during the first 3 1/2 months of the active phase of treatment if they are assigned to the CABA condition.
* Willingness to participate in audio-recorded sessions. (for treatment adherence)

Exclusion Criteria:

* Current diagnosis of moderate or severe substance (alcohol) use disorder using DSM-5 criteria within the past 30 days.
* Individuals with other psychiatric diagnoses will not be excluded except for bipolar disorder and psychotic disorders (requirement to refrain from additional treatments might be harmful).
* Veterans with a history indicated by medical record review of a diagnosis of moderate, severe, or penetrating TBI, or self-reported history on the Structured Interview for Collecting Head Trauma Event Characteristics of TBI with Post-Traumatic Amnesia (PTA) greater than 24 hours or loss of consciousness (LOC) greater than 30 minutes.
* Active suicidal intent indicating significant clinical risk, which would suggest that a treatment specifically targeting this intent was indicated. Clients who report suicidal ideation without imminent risk will be admitted into the study.
* Initiated psychotropic medication, including Prazosin, within 4 weeks or changed dosage within 2 weeks prior to the first assessment, as this would make it difficult to determine which treatment contributed to change in the CABA condition; additionally, started or changed dosage of sleep medication or low dosages of tricyclic antidepressant or trazodone for pain or sleep within 1 week prior to the first assessment. Participants could be reconsidered for eligibility after stability on medication was achieved. Enrollees will be asked to hold the doses of the current medications stable over the course of enrollment (though changes in medications after enrollment will not exclude them from on-going participation).
* Auditory or visual impairments that would compromise ability to participate or benefit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Callahan, PsyD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (2):
- United States (2):
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment as Usual (TAU): Treatment as Usual (TAU) is the usual care that patients would normally receive at the VA. TAU care involves psychotherapy (counseling) provided by a specialist in the treatment of PTSD. Patients will be offered individual appointments with an experienced provider on the PTSD Clinical Team (PCT). Beyond this, the specific approach will be determined by the patient and his/her provider and may include skills for managing PTSD and/or a chance for the patient to "process" his/her traumatic experiences. Additional treatments may be offered to patients. TAU may also include additional evaluation and/or treatment of mTBI. Treatment for mTBI includes individual or group sessions, and is based on clinical need.
  Treatment as Usual: TAU care involves psychotherapy (counseling) provided by a specialist in the treatment of PTSD. Patients will be offered individual appointments with an experienced provider on the PTSD Clinical Team (PCT). Beyond this, the specific approach will be determined by the patient and his/her provider and may include skills for managing PTSD and/or a chance for the patient to "process" his/her traumatic experiences. Additional treatments may be offered to patients, such as group classes and medications. TAU care may also include additional evaluation and/or treatment of mTBI, provided by the usual care offered in Portland or Seattle's respective neuropsychology clinics. Treatment for mTBI includes individual or group sessions, and is based on clinical need.
Period: Overall Study
Arm/Group | CABA | Treatment as Usual (TAU)
Started | 39 | 34
Completed | 30 | 26
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CABA | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 39 | 34 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 34 | 73
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 29 | 31 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 30 | 24 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 34 | 73
Years of Education [Mean (Standard Deviation); unit: years] | 14.58 (2.34) | 13.73 (1.99) | 14.19 (2.22)
Branch of Military Service [Count of Participants; unit: Participants]
  Army | 24 | 18 | 42
  Marines | 9 | 6 | 15
  Navy | 4 | 4 | 8
  Air Force | 2 | 3 | 5
  Coast Guard | 0 | 1 | 1
  Unreported | 0 | 2 | 2
Occupation Status [Count of Participants; unit: Participants]
  Employed | 19 | 15 | 34
  Unemployed | 20 | 19 | 39
Service Connection [Count of Participants; unit: Participants]
  Yes | 4 | 5 | 9
  No | 34 | 26 | 60
  Unreported | 1 | 3 | 4
Number of Deployments [Mean (Standard Deviation); unit: number of deployments] | 1.90 (1.01) | 2.24 (1.44) | 2.05 (1.22)

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptoms From Baseline as Measured by the Clinician Administered PTSD Scale - 5
Description: The Clinician Administered PTSD Scale (CAPS-IV; Blake et al., 1995; Weathers, Keane, & Davidson, 2001) was used to assess initial PTSD diagnosis (DSM-IV; APA, 2000) and PTSD symptom severity across assessment time points. The CAPS is considered a "gold standard" for assessing PTSD. Items are ranked on Likert scales according to both frequency (0-4) and intensity of symptoms (0-4), yielding an overall severity score based on the sum of frequency and intensity ratings across 17 items (range 0-136) . For this study, a diagnosis of PTSD was based on a scoring rule for items to be considered present of at least a "1" on frequency and "2" on intensity, with an overall severity score of at least 45 (Weathers, Ruscio, & Keane, 1999).
Time Frame: 0 weeks
Population: The total number of participants analyzed at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 39 | 34
score on a scale | 40.62 (10.65) | 40.53 (10.31)

2. Primary Outcome: PTSD Symptoms at 14 Weeks as Measured by the Clinician Administered PTSD Scale - 5
Description: as for outcome 1
Time Frame: 14 weeks
Population: The total number of participants analyzed is less than the total number of study participants due to incomplete or missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 25 | 23
score on a scale | 33.32 (13.43) | 37.35 (13.71)

3. Primary Outcome: PTSD Symptoms From Baseline as Measured by the PTSD Checklist-5
Description: The Posttraumatic Stress Disorder Checklist-Fifth Edition (PCL-5; Blanchard, Jones-Alexander, Buckley, & Forneris, 1996; Weathers, Litz, Herman, Huska, & Keane, 1993; Weathers et al., 2013) was used to assess participants subjective PTSD related distress. The PCL-5 is a 20 item self-report measure that assesses the presence of DSM-5 PTSD symptoms. Items are rated on a 5-point Likert scale ranging from 0 to 4 according to how much the symptom bothered the respondent over the past month. Total scores with scores range from 0-80, with higher scores indicating more symptomatic distress. Scores totaling 31 or more are associated with presumptive PTSD among military populations.
Time Frame: 0 weeks
Population: The total number of participants analyzed at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 39 | 34
score on a scale | 50.15 (14.48) | 51.21 (13.49)

4. Primary Outcome: PTSD Symptoms at 14 Weeks as Measured by the PTSD Checklist-5
Description: as for outcome 3
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 25 | 24
score on a scale | 44.92 (16.45) | 52.17 (16.66)

5. Primary Outcome: Baseline Memory as Measured by the Hopkins Verbal Memory Test - Revised
Description: The Hopkins Verbal Memory Test-Revised (HVLT-R; Brandt, 1991) is a measure of uncontextualized verbal learning and delayed recall. This score is converted to a standardized T-score (mean =50, S =10). The lower the T-score, the worse the performance.
Time Frame: 0 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 37 | 27
T-score | 35.05 (11.40) | 33.74 (10.84)

6. Primary Outcome: Memory at 14 Weeks as Measured by the Hopkins Verbal Memory Test - Revised
Description: as for outcome 5
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 20
T-score | 45.33 (13.58) | 37.30 (13.22)

7. Primary Outcome: Attention and Working Memory From Baseline as Measured by the Wechsler Adult Intelligence Scale-4th Edition, Digit Span Subtest
Description: The Wechsler Adult Intelligence Scale-4th Edition, Digit Span subtest (WAIS-IV; Wechsler, D., 2008) is a measure of attention and working memory. A higher total score indicates a higher level of performance (range 0-48). Raw scores are converted to scaled scores (e.g., 1-20), with higher scaled scores indicating a higher level of performance.
Time Frame: 0 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scaled score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 37 | 27
scaled score | 8.95 (2.52) | 9.22 (2.83)

8. Primary Outcome: Attention and Working Memory at 14 Weeks as Measured by the Wechsler Adult Intelligence Scale-4th Edition, Digit Span Subtest
Description: as for outcome 7
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scaled score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 20
scaled score | 10.46 (2.43) | 9.40 (2.87)

9. Primary Outcome: Verbal Fluency From Baseline as Measured by the Controlled Oral Word Association Test
Description: The Controlled Oral Word Association Test (COWAT; Ruff et al., 1996; Spreen, 1998) is a commonly used phonemic and semantic fluency word production test. A higher score indicates a higher level of performance (range 0-patient maximum).
Time Frame: 0 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 37 | 26
raw score | 43.68 (8.18) | 43.54 (11.93)

10. Primary Outcome: Verbal Fluency at 14 Weeks as Measured by the Controlled Oral Word Association Test
Description: as for outcome 9
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 20
raw score | 44.92 (7.52) | 41.05 (11.30)

11. Primary Outcome: Delis-Kaplan Executive Functions Scale (DKEFS) - Trails Subtest at Baseline
Description: The Delis-Kaplan Executive Function System, Trail Making subtest (D-KEFS; Delis, Kaplan, & Kramer, 2001; Delis, Kramer, Kaplan, & Holdnack, 2004) is a visual-motor task used to measure flexibility in thinking (executive function) and processing speed. Raw scores are converted to scaled scores (e.g., 1-20). A higher score indicates a higher level of performance. This scale is measuring Trial 4.
Time Frame: 0 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scaled score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 36 | 27
scaled score | 9.08 (3.68) | 8.30 (3.58)

12. Primary Outcome: Processing Speed at 14 Weeks as Measured by Delis-Kaplan Executive Functions Scale (DKEFS) Trails Subtest
Description: as for outcome 11
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scaled score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 23 | 19
scaled score | 10.61 (3.09) | 9.79 (2.53)

13. Secondary Outcome: Symptoms of Depression From Baseline as Measured by the Beck Depression Inventory -II
Description: The Beck Depression Inventory-II (BDI-II; Beck, Steer, & Brown, 1996) is a 21-item measure of subjective levels of depression. Items are rated on a 3-point Likert scale with higher scores reflecting greater severity of symptoms (range 0-63).
Time Frame: 0 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 39 | 33
raw score | 29.74 (12.02) | 30.10 (9.62)

14. Secondary Outcome: Symptoms of Depression at 14 Weeks as Measured by the Beck Depression Inventory -II
Description: as for outcome 13
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 25 | 24
raw score | 24.96 (13.26) | 31.17 (11.41)

15. Secondary Outcome: Global Life Satisfaction From Baseline as Measured by the Satisfaction With Life Scale
Description: The Satisfaction with Life Scale (SWLS; Diener, Emmons, Larsen, & Griffin, 1985) is a brief measure of global life satisfaction or quality of life. Items are rated on a 7-point Likert scale with higher scores indicating greater satisfaction (range 5-35).
Time Frame: 0 weeks
Population: The total number of participants analyzed at baseline.
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 39 | 34
raw score | 15.38 (6.37) | 15.41 (7.72)

16. Secondary Outcome: Global Life Satisfaction at 14 Weeks as Measured by the Satisfaction With Life Scale
Description: as for outcome 15
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 25 | 22
raw score | 16.92 (7.39) | 15.32 (8.07)

17. Secondary Outcome: Postconcussion Symptoms From Baseline as Measured by the Neurobehavioral Symptom Inventory
Description: The Neurobehavioral Symptom Inventory (NSI; Cicerone, K.D. & Kalmer, K., 1995) is a post-concussive symptom measure recommended for use in military studies. Items are rated on a 4-point Likert scale with higher scores reflecting greater severity of symptom disturbance since time of injury (range 0-66).
Time Frame: 0 weeks
Population: The total number of participants analyzed at baseline.
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 39 | 34
raw score | 45.79 (14.81) | 46.38 (10.96)

18. Secondary Outcome: Postconcussion Symptoms at 14 Weeks as Measured by the Neurobehavioral Symptom Inventory
Description: as for outcome 17
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 25 | 23
raw score | 42.72 (17.51) | 49.43 (14.88)

19. Secondary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: The CSQ is an 8-item questionnaire rated on a Likert scale of 1-4 used to assess client's treatment satisfaction. Scores range from 8-32, with higher scores equaling greater satisfaction.
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Groups:
- Treatment as Usual (TAU): Treatment as Usual (TAU) is the usual care that patients would normally receive at the VA. TAU care involves psychotherapy (counseling) provided by a specialist in the treatment of PTSD. Patients will be offered individual appointments with an experienced provider on the PTSD Clinical Team (PCT). Beyond this, the specific approach will be determined by the patient and his/her provider and may include skills for managing PTSD and/or a chance for the patient to "process" his/her traumatic experiences. Additional treatments may be offered to patients. TAU may also include additional evaluation and/or treatment of mTBI. Treatment for mTBI includes individual or group sessions, and is based on clinical need.
  Treatment as Usual: TAU care involves psychotherapy (counseling) provided by a specialist in the treatment of PTSD. Patients will be offered individual appointments with an experienced provider on the PTSD Clinical Team (PCT). Beyond this, the specific approach will be determined by the patient and his/her provider and may include skills for managing PTSD and/or a chance for the patient to "process" his/her traumatic experiences. Additional treatments may be offered to patients, such as group classes and medications. TAU care may also include additional evaluation and/or treatment of mTBI. Treatment for mTBI includes individual or group sessions, and is based on clinical need.
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 21
raw score | 27.75 (6.07) | 27.24 (3.29)

20. Other Pre Specified Outcome: Use of Cognitive Strategies From Baseline as Measured by the Memory Compensation Questionnaire
Description: Memory Compensation Questionnaire (MCQ)70. Rates the extent to which patients use various strategies to improve memory performance. 44 Items are rated on a 5-point Likert scale with higher scores indicating grater use of compensatory strategies (range 0-176).
Time Frame: 0 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 38 | 33
raw score | 120.18 (28.67) | 120.97 (28.46)

21. Other Pre Specified Outcome: Use of Cognitive Strategies at 14 Weeks as Measured by the Memory Compensation Questionnaire
Description: as for outcome 20
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 20
raw score | 121.38 (25.80) | 115.55 (45.06)

22. Other Pre Specified Outcome: Postconcussion Symptoms From Baseline as Measured by the Rivermead Postconcussive Questionnaire
Description: Rivermead Post Concussive Symptom Questionnaire (RPQ) will be used to measure postconcussive symptoms. Items are rated on a 5-point Likert scale with a higher number indicating more severe PCS (range 0-64).
Time Frame: 0 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 38 | 33
raw score | 40.76 (12.39) | 39.45 (12.03)

23. Other Pre Specified Outcome: Postconcussion Symptoms at 14 Weeks as Measured by the Rivermead Postconcussive Questionnaire
Description: as for outcome 22
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 21
raw score | 35.35 (15.44) | 37.42 (15.07)

24. Other Pre Specified Outcome: Symptoms of Anxiety From Baseline as Measured by the Brief Symptom Inventory
Description: Brief Symptom Inventory 18 (BSI 18) is a measure of anxiety symptoms. 18 items are rated on a 5-point Likert scale with higher scores indicating more severe symptoms (range 0-72).
Time Frame: 0 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 38 | 32
raw score | 30.87 (14.33) | 30.91 (13.72)

25. Other Pre Specified Outcome: Symptoms of Anxiety at 14 Weeks as Measured by the Brief Symptom Inventory
Description: as for outcome 24
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 22
raw score | 26.54 (15.49) | 29.56 (15.76)

26. Other Pre Specified Outcome: Health Related Quality of Life From Baseline as Measured by the Neuro-Quality of Life Satisfaction With Social Roles and Activities.
Description: Neuro-QOL Satisfaction with Social Roles and Activities is a health-related quality of life assessment tool. Eight items are rated on a 5-point Likert scale. Scores were converted to T-scores (mean = 50; SD = 10). Lower T-scores indicate greater dissatisfaction.
Time Frame: 0 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 38 | 32
T-score | 38.37 (8.06) | 32.38 (15.41)

27. Other Pre Specified Outcome: Health Related Quality of Life at 14 Weeks as Measured by the Neuro-Quality of Life Satisfaction With Social Roles and Activities.
Description: as for outcome 26
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 22
T-score | 37.90 (12.82) | 38.72 (4.80)

28. Other Pre Specified Outcome: Functional Impairment From Baseline as Measured by the Sheehan Disability Scale
Description: The Sheehan Disability Scale is a brief self-report measure of functional impairment across three primary life domains: work/school, social life, and family life/home responsibilities. Participants rated how much their symptoms bothered or distress them over the past week on a scale from 0 (not at all) to 10 (extremely), with higher scores indicating greater functional impairment. Total scores (possible range 0-30) were used in analyses.
Time Frame: 0 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 36 | 33
raw score | 20.06 (7.43) | 21.50 (6.06)

29. Other Pre Specified Outcome: Functional Impairment at 14 Weeks as Measured by the Sheehan Disability Scale
Description: as for outcome 28
Time Frame: 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CABA | Treatment as Usual (TAU)
Number analyzed (Participants) | 21 | 22
raw score | 15.57 (7.77) | 18.36 (8.33)

ADVERSE EVENTS:
Time Frame: Baseline to 6-month follow up. AEs were documented at baseline, 7 weeks, 14 weeks, and 39 weeks, or in between visits if study staff were alerted to an event during treatment.
Arm/Group | CABA | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/39 | 0/34
Other Adverse Events (participants affected / at risk) | 3/39 | 3/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CABA (N=39) | Treatment as Usual (TAU) (N=34)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0) — Patient had a panic attack during the session. She was walked to the ED and discharged a short time later.
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) — Participant taken to ED due to SI with vague plan.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CABA (N=39) | Treatment as Usual (TAU) (N=34)
Passive SI (Psychiatric disorders) | 2 (2) | 0 (0)
Emergency Department Visit (General disorders) | 1 (2) | 3 (5) — injury/pain

LIMITATIONS AND CAVEATS:
This study experienced significant recruitment delays and difficulties associated with delayed IRB approvals and COVID-era shutdowns. As a result, the sample size is smaller than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT02391402/Prot_SAP_000.pdf